CLINICAL TRIAL: NCT06401824
Title: A Single Arm Phase II Study Evaluating Intracranial Efficacy of Sacituzumab Govitecan (SG) With Bevacizumab in Patients With Active, Asymptomatic Brain Metastases From Non-small Cell Lung Cancer (NSCLC)
Brief Title: Sacituzumab Govitecan and Bevacizumab for NSCLC Brain Metastases
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CO-NL-979-6888
Record Dates: First submitted 2024-05-02; First posted 2024-05-07 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: NSCLC Stage IV; Brain Metastases, Adult
Keywords: non small cell lung cancer; brain metastases; bevacizumab; sacituzumab govitecan
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Brain Neoplasms | interventions — Bevacizumab; sacituzumab govitecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- sacituzumab govitecan (SG) plus bevacizumab (Experimental): SG 10mg/kg intravenous day 1 and day 8 of a 21-day cycle, + bevacizumab 15 mg/kg iv day 1 of a 21-day cycle till unacceptable toxicity or disease progression.
  Interventions: Drug: Sacituzumab Govitecan-Hziy 180 MG plus bevacizumab

INTERVENTIONS:
Drug: Sacituzumab Govitecan-Hziy 180 MG plus bevacizumab — Sacituzumab govitecan 10mg/kg intravenous day 1 and day 8 of a 21-day cycle, + bevacizumab 15 mg/kg iv day 1 of a 21-day cycle till unacceptable toxicity or disease progression.
  Other Names: sacituzumab govitecan; zirabev

SUMMARY:
This study will evaluate whether the combination of sacituzumab govitecan (SG) and bevacizumab will result in shrinkage of brain metastases from patients with non-squamous non-small cell lung cancer (NSCLC), with disease progression on chemotherapy and immunotherapy.

DETAILED DESCRIPTION:
Historically, the prognosis for patients with non-small cell lung cancer (NSCLC) brain metastases (BM) was poor, but this paradigm is slowly shifting as current data with an immune checkpoint inhibitor (ICI) based regimen show that a subgroup of patients with BM can achieve long-term survival. For patients with disease progression in the brain after platinum-doublet chemotherapy and ICI, no good systemic treatment options exist and due to local treatments, systemic therapy is often delayed. Of note, most of these patients also have extra-cranial disease progression which needs to be treated. The current standard of care post chemo-ICI progression is docetaxel, with dismal outcomes. The same holds true for patients with NSCLC with an actionable genomic alteration. Upon exhaustion of targeted therapies and platinum-doublet chemotherapy with or without ICI, the standard of care is docetaxel with the same dismal outcomes. Therefore, new systemic therapies that are active systemically as well as intracranially are needed in this population. Antibody-drug-conjugates (ADC) are promising new drugs and several have entered testing in randomized phase III trials. In the majority of the trials evaluating ADCs, patients with untreated BM were excluded. Importantly, Sacituzumab Govitecan (SG), a TROP2-ADC, achieves therapeutic concentrations of SN-38, the active payload of SG, in the CNS. SG is evaluated versus docetaxel in the ongoing EVOKE-1 trial (NCT05089734) but patients with untreated BM are excluded. Preclinically, SG combined with bevacizumab, but not with cetuximab, significantly improved survival over SG alone. Bevacizumab combined with chemotherapy results in an impressive intracranial ORR of 61%. Of note, a possible pseudo response (a marked decrease in contrast enhancement and oedema on MR imaging that often occurs after the initiation of bevacizumab therapy, attributed to normalization of the blood-brain barrier), was not taken into account. Pharmacokinetic drug-drug interactions between bevacizumab and SG are not expected given the distinct proteolytic catabolism responsible for degradation of each monoclonal antibody (moiety). In addition, SN-38 is metabolized by UGT1A1, which is not affected by bevacizumab. Based on the data above, it is of interest to also evaluate SG combined with bevacizumab in patients with BM from NSCLC. This will be evaluated in patients with non-squamous non-small cell lung cancer (NSCLC), with disease progression on chemotherapy and immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

* In order to be eligible to participate in this study, a subject must meet all of the following criteria:

  1. Signed informed consent must be obtained prior to participation in the study.
  2. Participant is an adult ≥ 18 years of age at the time of informed consent.
  3. ECOG performance status ≤1.
  4. Estimated life expectancy of 12 weeks or more.
  5. Pathology proven metastatic non-squamous NSCLC
  6. For those without an actionable oncogenic driver: progression on immunotherapy and/or platinum-doublet chemotherapy (concurrent or sequential, in any order). If contra-indication for immunotherapy: progression on platinum-doublet chemotherapy.
  7. For those with an actionable oncogenic driver: progression on targeted therapy and platinum-doublet chemotherapy. For the latter group, previous ICI is allowed but not mandatory.
  8. BM not in eloquent area (all patients have at least to be discussed with a neurologist, and preferably they are discussed in the local neuro-oncology MDT).
  9. Maximum BM size 2 cm in longest diameter (for each BM).
  10. At least one untreated brain metastasis ≥ 5mm:

      1. Patients with largest measurable intracranial lesion ≥5 mm but <10 mm may be allowed to enroll upon agreement with the principal investigator (for patients with target lesions of ≥ 5mm but <10 mm, 1.5 mm slice thickness brain MRI is required).
      2. Prior local treatment is permissible provided unequivocal progression in the lesion has since occurred (discussed in neuro-oncology MDT) or if new lesions have occurred.
      3. For at least 7 days prior to first dose of SG and bevacizumab in this study: Patient must be asymptomatic from CNS metastases and on a stable dose of corticosteroids, with a maximum of 4 mg dexamethasone/day. Anti-epileptic dose should also be stable for 7 days.
  11. Participant must have recovered from all toxicities related to prior treatments to grade ≤ 1 (CTCAE v 5.0). Exception to this criterion are alopecia and neuropathy of any grades.
  12. Adequate organ function including the following laboratory values at the screening visit:

      * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L (without growth factor support),
      * Platelets ≥ 100 x 109/L (without growth factor support),
      * Hemoglobin (Hb) ≥ 6 mmol/l (= 9 g/dl) (7 days without transfusions or growth factor support),
      * Aspartate transaminase (AST) ≤ 2.5 x ULN, or ≤ 5 × ULN if known liver metastases
      * Alanine transaminase (ALT) ≤ 2.5 x ULN, or ≤ 5 × ULN if known liver metastases
      * Serum albumin > 3 g/dL
      * Total bilirubin ≤ 1.5 ULN,
      * Creatinine clearance ≥ 30 mL/min by calculation using Cockcroft-Gault formula or based on 24-hour urine sample assessment.
  13. Participant is capable of following instructions regarding study treatment administration, and must be able to communicate with the Investigator and comply with the requirements of the study procedures.
  14. Negative serum or urine pregnancy test within 7 days prior to study treatment in women with childbearing potential. Patient must be willing to use effective methods of contraception. Female patients must be postmenopausal, surgically sterile, or they must agree to use a physical barrier method of contraception in addition to either an intrauterine device or hormonal contraception until at least 4 months after termination of study drug.

Exclusion Criteria:

* A potential subject who meets any of the following criteria will be excluded from participation in this study:

  1. Leptomeningeal metastasis (based on MRI or CSF cytology, if strong suspicion despite negative MRI, CSF analysis should be done).
  2. Previous treatment with TROP2 inhibitor or angiogenesis inhibitor.
  3. Known hypersensitivity to the study drugs, its metabolites, or formulation excipient.
  4. Positive serum pregnancy test or women who are breastfeeding.
  5. Contra-indication for MRI.
  6. History of allogeneic bone marrow or solid organ transplant.
  7. Have had a prior anticancer biologic agent (ADC, ICI) within 4 weeks prior to enrolment or have had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to enrolment and have not recovered (ie, ≥ Grade 2 is considered not recovered) from AEs at the time of study entry.

     a. Note: Patients participating in observational studies are eligible.
  8. Have not recovered (ie, ≥ Grade 2 is considered not recovered) from AEs due to a previously administered agent.

     1. Note: patients with any grade vitiligo or alopecia are an exception to this criterion and will qualify for the study.
     2. Note: if patients received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
  9. Have an active second malignancy. Note: patients with a history of malignancy that has been treated completely, with no evidence of active cancer for 3 years prior to enrollment, or patients with surgically cured tumours with low risk of recurrence (eg, nonmelanoma skin cancer, histologically confirmed complete excision of carcinoma in situ, or similar) are allowed to enroll.
  10. Met any of the following criteria for cardiac disease:

      1. Myocardial infarction or unstable angina pectoris within 6 months of enrollment.
      2. History of serious ventricular arrhythmia (ie, ventricular tachycardia or ventricular fibrillation), high-grade atrioventricular block, or other cardiac arrhythmias requiring antiarrhythmic medications (except for atrial fibrillation that is well controlled with antiarrhythmic medication); history of QT interval prolongation.
      3. New York Heart Association (NYHA) class III or greater congestive heart failure or left ventricular ejection fraction of < 40%.
  11. Have active chronic inflammatory bowel disease (ulcerative colitis, Crohn's disease) or GI perforation within 6 months of enrolment.
  12. Have active serious infection requiring antibiotics.
  13. Have known history of HIV-1 or 2 (or positive HIV-1/2 antibody, if done at screening) with detectable viral load OR taking medications that may interfere with SN-38 metabolism.
  14. Have known active hepatitis B virus (HBV) or hepatitis C virus (HCV). In patients with a history of HBV or HCV, patients with detectable viral loads will be excluded.
  15. Have other concurrent medical or psychiatric conditions that, in the investigator's opinion, may be likely to confound study interpretation or prevent completion of study procedures and follow-up examinations.
  16. Any medical condition that, in the investigator's or sponsor's opinion, poses an undue risk to the patient's participation in the study
  17. Use of other investigational drugs (drugs not marketed for any indication) within 28 days or 5 half-lives (whichever is longer) of first dose of study drug.
  18. Clinically severe pulmonary compromise resulting from intercurrent pulmonary illnesses including, but not limited to, any underlying pulmonary disorder (ie, pulmonary embolism within 1 months of enrolment, severe asthma, severe chronic obstructive pulmonary disease, restrictive lung disease, uncontrolled pleural effusion, etc.); any autoimmune, connective tissue, or inflammatory disorders with pulmonary involvement (ie, rheumatoid arthritis, Sjogren syndrome, sarcoidosis, etc.); or prior pneumonectomy.
  19. Contra-indications specific to bevacizumab

      1. Inadequately controlled hypertension (defined as systolic blood pressure > 150 mmHg and/or diastolic blood pressure > 100 mmHg). Anti-hypertensive therapy to achieve these parameters is allowable.
      2. Prior history of hypertensive crisis or hypertensive encephalopathy.
      3. Significant vascular disease (e.g., aortic aneurysm requiring surgical repair or recent peripheral arterial thrombosis) within 6 months prior to start of treatment.
      4. History of hemoptysis (≥ one-half teaspoon of bright red blood per episode) within 1 month prior to start of treatment.
      5. Evidence of bleeding diathesis or coagulopathy (in the absence of therapeutic anticoagulation).
      6. Current or recent (within 10 days of start of treatment) use of aspirin (> 325 mg/day) or treatment with dipyridamole, ticlopidine, clopidogrel, and cilostazol.
      7. Current use of full-dose oral or parenteral anticoagulants or thrombolytic agents for therapeutic purposes that has not been stable for > 2 weeks prior to start of treatment. The use of full-dose oral or parenteral anticoagulants is permitted as long as the INR or aPTT is within therapeutic limits (according to the medical standard of the enrolling institution) and the patient has been on a stable dose of anticoagulants for at least 2 weeks prior to start of treatment.
      8. Prophylactic anticoagulation for the patency of venous access devices is allowed, provided the activity of the agent results in an INR < 1.5 × ULN and aPTT is within normal limits within 14 days prior to start of treatment.
      9. Prophylactic use of low-molecular-weight heparin (i.e., enoxaparin 40 mg/day) is permitted.
      10. Core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 7 days prior to the first dose of bevacizumab.
      11. History of abdominal or tracheoesophageal fistula or gastrointestinal perforation within 6 months prior to start of treatment.
      12. Clinical signs of gastrointestinal obstruction or requirement for routine parenteral hydration, parenteral nutrition, or tube feeding.
      13. Evidence of abdominal free air not explained by paracentesis or recent surgical procedure.
      14. Serious, non-healing wound, active ulcer, or untreated bone fracture.
      15. Proteinuria, as demonstrated by urine dipstick or > 1.0 g of protein in a 24-hour urine collection. All patients with ≥ 2+ protein on dipstick urinalysis at baseline must undergo a 24-hour urine collection and must demonstrate ≤ 1 g of protein in 24 hours.
      16. Clear tumour infiltration into the thoracic great vessels is seen on imaging.
      17. Clear cavitation of pulmonary lesions is seen on imaging.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-04-24 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
brain metastases overall response rate (ORR) | up to 24 months
  ORR is defined as the proportion of patients with best overall response of complete response (CR) or partial response (PR) based on central and local investigator's assessment according to RANO-BM criteria on brain MRI

SECONDARY OUTCOMES:
brain metastases overall response rate (ORR) with correction for bevacizumab-pseudoresponse | up to 24 months
  ORR is defined as the proportion of patients with best overall response of complete response (CR) or partial response (PR) based on central and local investigator's assessment according to RANO-BM criteria on brain MRI with additional criteria for potential pseudo response due to bevacizumab
brain metastases disease control rate (DCR) | up to 24 months
  DCR is defined as the proportion of participants with Best Overall Response (BOR) of Complete Response (CR), Partial Response (PR), Stable Disease (SD) or Non-CR/Non-PD according to RANO-BM on brain MRI
CNS progression free survival (PFS) | up to 24 months
  PFS is the time from date of start of treatment to the date of event defined as the first documented progression or death due to any cause. PFS is based on local and central assessment according to RANO-BM on brain MRI
Extracranial ORR and DCR | up to 24 months
  ORR is defined as the proportion of patients with best overall response of complete response (CR) or partial response (PR) based on local investigator's assessment, DCR is defined as the proportion of participants with Best Overall Response (BOR) of Complete Response (CR), Partial Response (PR), Stable Disease (SD) or Non-CR/Non-PD according to RECIST 1.1, measured with CT
Extracranial PFS | up to 24 months
  PFS is the time from date of start of treatment to the date of event defined as the first documented progression or death due to any cause. PFS is based on local assessment according to RECIST 1.1 based on CT
overall PFS | up to 24 months
  median overall PFS based on RANO-BM for BM and RECIST 1.1 for extracranial lesions as defined above
overall survival | up to 33 months
  OS is defined as the time from date of start of treatment to date of death due to any cause
Safety according to CTCAE v5.0 | up to 33 months
  according to CTCAE v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Lizza Hendriks, MD, PhD, Principal Investigator — Maastricht University Medical Hospital
Locations (3):
- Netherlands (3):
  - NKI-AvL, Amsterdam
  - University Medical Center Groningen, Groningen
  - Maastricht University Medical Center, Maastricht

IPD SHARING:
Plan to Share IPD: No